CLINICAL TRIAL: NCT00615420
Title: A Randomized Placebo-Controlled Trial of Manuka Honey for Oral Mucositis Due to Radiation Therapy for Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: H07-02297; H07-02297
Record Dates: First submitted 2008-02-04; First posted 2008-02-14 (Estimated); Results first posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2012-05

CONDITIONS: Radiotherapy Induced Mucositis; Head and Neck Cancer
Keywords: Mucositis; Radiation; Honey
MeSH Terms: conditions — Head and Neck Neoplasms; Mucositis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study was blinded to all except necessary pharmacy staff until after the study was closed.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Manuka Honey (Experimental): Irradiated organic manuka honey 5ml 4 times a day held in mouth for 30 secs then swallowed
  Interventions: Dietary Supplement: manuka honey
- Placebo (Placebo Comparator): Sugar-free placebo gel 5ml 4 times a day, swished and held in mouth for 30 secs then swallowed
  Interventions: Dietary Supplement: placebo gel

INTERVENTIONS:
Dietary Supplement: manuka honey — Irradiated organic manuka honey 5ml 4 times a day held in mouth for 30 secs then swallowed. May be diluted with equal or twice the volume of water to reduce nausea in patients already nauseated from chemotherapy.
  Arms: Manuka Honey
Dietary Supplement: placebo gel — Sugar-free honey-flavoured gel 5ml 4 times a day swished and held in mouth for 30 secs then swallowed. May be diluted with equal or twice the volume of water to reduce nausea in patients already nauseated from chemotherapy.
  Arms: Placebo

SUMMARY:
The primary hypothesis of this study is that regular topical oral application of Manuka Honey will reduce the severity and duration of oral mucositis in patients who are undergoing mucotoxic radiation therapy for cancer treatment.

DETAILED DESCRIPTION:
Oral mucositis is a common side-effect of radiation therapy for many head and neck cancers, and can have a very severe impact on quality of life and nutritional status. At least42% of patients treated for head and neck cancers will develop grade 3 or 4 oral mucositis. Although there have been positive trials, no study has had overwhelming data to strongly support any one agent in the prevention or treatment of oral mucositis. A comprehensive review of the literature done in 2004 found only benzydamine (a topical nonsteroidal anti-inflammatory agent) to be beneficial as a palliative treatment for established mucositis. Management essentially consists of pain management, with topical and oral analgesics/anaesthetics and anti-inflammatory agents, and nutritional support, once mucositis is established. Despite the use of these agents, many patients still have severe mucositis, and there is great need for new treatments to reduce this distressing complication of cancer therapy.

Currently, the only standard "treatment" consists of an oral rinse of warm water, salt, and baking soda 4 times a day. This is only to maintain oral hygiene and does not have any impact on the severity or duration of the mucositis itself. Topical fluoride is applied at bedtime to reduce the caries risk. Basic oral care (brushing and flossing as tolerated) is recommended to maintain general mucosal health and to reduce the impact of oral microbial flora.

Study Objectives The primary objective of this study is to see if topical oral Manuka honey reduces the severity of mucositis in patients receiving radiation treatment for head and neck cancer. Secondary objectives are to assess the impact of any demonstrated improvement in mucositis on nutrition, symptom burden, quality of life, and radiotherapy treatment interruptions.

ELIGIBILITY:
Inclusion Criteria:

* Patients commencing radiation therapy of 50 Gy or higher with the dosage field affecting the oral mucosa unilaterally or bilaterally (minimum 3 observable sites affected).
* Patients willing and able to attend weekly assessments throughout their treatment, plus one week after completion of treatment.

Exclusion Criteria:

* Patients unable to understand the consent process (translators will be used if necessary so being English-speaking is not required).
* Patients unable to attend the follow-up visits
* Patients participating in other clinical trials which might affect the severity of mucositis
* Patients allergic to honey, multiple pollens, or to celery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-07; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippa Hawley, B.Med, Principal Investigator — British Columbia Cancer Agency
Locations (2):
- Canada (2):
  - BC Cancer Agency, Surrey, British Columbia
  - BC Cancer Agency, Vancouver, British Columbia

RESULTS

PARTICIPANT FLOW:
Groups:
- Honey: Irradiated organic manuka honey 5ml 4 times a day held in mouth for 30 secs then swallowed
  manuka honey: Irradiated organic manuka honey 5ml 4 times a day held in mouth for 30 secs then swallowed. May be diluted with equal or twice the volume of water to reduce nausea in patients already nauseated from chemotherapy.
Period: Overall Study
Arm/Group | Honey | Placebo
Started | 54 | 52
Completed | 23 | 25
Not Completed | 31 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Honey | Placebo | Total
Number analyzed (Participants) | 54 | 52 | 106
Age, Continuous [Mean (Full Range); unit: years] — Population: Not all patients have baseline information available
  years
    number analyzed (Participants) | 52 | 48 | 100
    (all) | 56.8 [32 to 100] | 59.5 [41 to 85] | 58.1 [32 to 100]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Not all patients have baseline information available
  Participants
    number analyzed (Participants) | 54 | 50 | 104
    Female | 10 | 8 | 18
    Male | 44 | 42 | 86
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Weight [Mean (Standard Deviation); unit: kg] — Population: Not all patients have baseline information available
  kg
    number analyzed (Participants) | 52 | 50 | 102
    (all) | 85.6 (19.3) | 79.6 (15.2) | 82.7 (17.6)
Diabetic [Count of Participants; unit: Participants] | 3 | 10 | 13
Smoker [Count of Participants; unit: Participants] | 9 | 7 | 16
ECOG > 0 [Count of Participants; unit: Participants] | 8 | 13 | 21
Chemotherapy [Count of Participants; unit: Participants] | 31 | 35 | 66
Radiation Therapy => 7,000 Gy [Count of Participants; unit: Participants] — Gy = Gray; the international system unit of radiation dose
  Participants | 36 | 30 | 66

OUTCOME MEASURES:

1. Primary Outcome: Severity of Mucositis According to the Radiation Therapy Oncology Group (RTOG) for Patients Who Had at Least One Mucositis Assessment
Description: Worst Radiation Therapy Oncology Group (RTOG) score greater than or equal to Grade 3 mucositis The scale ranges from Grade 0 (No mucositis) to Grade 4 (Necrosis or deep ulceration ± bleeding) where Grade 0 is the best outcome and Grade 4 is the worst outcome.
Time Frame: Over 7 weeks of expected duration of mucositis
Population: Patients who had at least one mucositis assessment were included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Honey | Placebo
Number analyzed (Participants) | 40 | 41
Participants | 14 | 18

2. Primary Outcome: Severity of Mucositis According to the Radiation Therapy Oncology Group (RTOG) for Patients Who Had a Minimum of 2 Mucositis Assessments
Description: as for outcome 1
Time Frame: Over 7 weeks of expected duration of mucositis
Population: Patients who had a minimum of 2 mucositis assessments were included in this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Honey | Placebo
Number analyzed (Participants) | 31 | 33
Participants | 11 | 16

ADVERSE EVENTS:
Arm/Group | Honey | Placebo
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/52
Other Adverse Events (participants affected / at risk) | 8/54 | 6/52
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Honey (N=54) | Placebo (N=52)
Nausea (Gastrointestinal disorders) | 8 | 5
Bad Taste (Product Issues) | 0 | 1
Burning Sensation in Mouth (Product Issues) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No